CLINICAL TRIAL: NCT00519701
Title: Effects of Hydroxyurea on the Prevention of Chronic Organ Damage in Young Children With Sickle Cell Anemia
Brief Title: Hydroxyurea in Young Children With Sickle Cell Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3297
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Sickle Cell Anemia
Keywords: sickle cell anemia; hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): hydroxyurea
  Interventions: Drug: hydroxyurea

INTERVENTIONS:
Drug: hydroxyurea

SUMMARY:
The purpose of this study is to asses prospectively the safety and efficacy of hydroxyurea therapy in children with Sickle cell Anemia between ages 18 months and 5 years, with special emphasis on the ability of hydroxyurea to prevent or reverse chronic organ damage.

DETAILED DESCRIPTION:
Previous studies have shown that hydroxyurea therapy in adults and older children with SCA improves laboratory parameters and ameliorates the clinical severity of disease. Little is known, however, about the effects of hydroxyurea on the chronic organ damage that occurs in patients with SCA and leads to significant morbidity and mortality in young adults. The objectives of this study are to assess the safety and efficacy of HU in young children with SCA and to determine whether HU preserves renal function, reduces transcranial doppler ultrasound (TCD) values, and prevents development of brain ischemia as evidenced by MRI/MRA imaging. In addition, we will evaluate the effects of hydroxyurea on quality of life

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Sickle Cell Anemia (Hb SS or Hb S beta zero-thalassemia)

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2002-04; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Transcranial doppler ultrasound velocity | 2 years
Magnetic resonance imaging/angiography | 2 years
Glomerular Filtration Rate | 2 years
Quality of Life | 2 years
Neurocognitive outcomes | 2 years

SECONDARY OUTCOMES:
Growth parameters | 2 years
Hematological parameters | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Thornburg, MD mS, Principal Investigator — Duke University
Locations (1):
- Duke University Medican Center, Durham, North Carolina, United States